CLINICAL TRIAL: NCT04262440
Title: The Effect of Caloric Supplement in the Clinical Outcomes in Acute Lung Injury Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Wang, Chen-Yu, Director of Medical ICU, Taichung Veterans General Hospital
Other Study IDs: CF19068A
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: ARDS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The optimal amount caloric intake were still controversy in critically ill patients in literature. There were no significant outcome difference with different caloric intake in acute lung injury patients. In order to identify the optimal amount caloric intake in acute lung injury patients, we conduct a prospectively observational study to see whether the caloric differences influence hospital mortality.

DETAILED DESCRIPTION:
The is a prospectively observational study. The data including basic demographic data, daily PN/EN caloric intake, days of ICU stay, days of hospital stay, hospital mortality, days of ventilator use.. will be collected. Statistic analysis included chi-square, student t test, logistic regression and ROC curve will be applied to analyze the different characteristics between survived and died patients. Also we can figure out the optimal cut value of caloric intake with best outcome by ROC curve analysis. We plan enrolled 200 participants within study period.

ELIGIBILITY:
Inclusion Criteria:

Age older than 20 year old Respiratory failure with ventilator Fit the diagnostic criteria of ARDS (2012 Berlin Criteria)

Exclusion Criteria:

Expected ICU stay less than 72 hours

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age older than 20 year old Respiratory failure with ventilator Fit the diagnostic criteria of ARDS
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: CHEN-YU WANG, MHA, Principal Investigator — Department of Critical Care Medicine, Taichung Veterans General hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, 台中市, Taiwan